CLINICAL TRIAL: NCT04067128
Title: Pilot of Brief Health Coaching Intervention to Improve Adherence to Positive Airway Pressure Therapy: Retroactive Analysis of a Quality Improvement Project
Brief Title: Health Coaching for Positive Airway Pressure Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Rachel Willard-Grace, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-23281
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to receive health coaching or usual care. For the health coaching arm, an unlicensed, trained health coach called patients three times to identify and resolve barriers to adherence, including lack of understanding of their condition or the treatment, discomfort in acclimating to treatment, technical difficulties in mask fit or device settings, and challenges in navigating durable medical equipment providers. Patients assigned to usual care had access to all other available resources, including technical support from durable medical equipment providers, respiratory therapist visits with the Sleep Clinic, group visits, or visits with their primary care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health coaching arm (Experimental): For the health coaching arm, an unlicensed, trained health coach called patients three times to identify and resolve barriers to adherence, including lack of understanding of their condition or the treatment, discomfort in acclimating to treatment, technical difficulties in mask fit or device settings, and challenges in navigating durable medical equipment providers.
  Interventions: Behavioral: Health coaching
- Usual care arm (No Intervention): Patients assigned to usual care had access to all other available resources, including technical support from durable medical equipment providers, respiratory therapist visits with the Sleep Clinic, group visits, or visits with their primary care provider.

INTERVENTIONS:
Behavioral: Health coaching — Brief telephonic intervention consisting of up to three phone calls
  Arms: Health coaching arm

SUMMARY:
This study tested a low-resource, brief telephonic health coaching intervention to improve adherence to positive airway pressure therapy for treatment of sleep apnea.

DETAILED DESCRIPTION:
We conducted post hoc analysis of a quality improvement initiative in which patients were randomly assigned to receive health coaching or usual care. Participants were English- and Spanish-speaking patients from a county-based public health system who had previously received a positive airway pressure device for the treatment of sleep apnea. An unlicensed, trained health coach called patients three times to resolve barriers to adherence. Adherence measures collected by device modem at baseline and 4 weeks were the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* At least 18 years of age
* Had previously received a modem-enabled positive airway pressure device for the treatment of sleep apnea
* Received care from the San Francisco General Hospital Sleep Clinic

Exclusion Criteria:

* Not English- or Spanish-speaking
* Younger than 18 years
* Does not have phone number at which could be reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion using device at any time in last 30 days | Enrollment to 30 days post enrollment
  Numerator: Number of people using device at any time in last 30 days; Denominator: Number of people in study arm

SECONDARY OUTCOMES:
Mean number of hours used on average over the last 30 days | Enrollment to 30 days post enrollment
  Total number of hours device used during 30 day period divided by 30 days
Mean number of hours used on average over the last 30 days on nights that device was used | Enrollment to 30 days post enrollment
  Total number of hours device used during 30 day period divided by the number of days on which the device was used
Mean proportion of last 30 days in which device used at least 4 hours/night | Enrollment to 30 days post enrollment
  Mean across group of: (Numerator: Number of days in last 30 days that device was used at least 4 hours; Denominator: 30 days)
Proportion meeting Medicare standard for adherence (at least 4 hours/night for at least 70% of last 30 days) | Enrollment to 30 days post enrollment
  Numerator: Number of people meeting Medicare standard for adherence; Denominator: Number of people in study arm

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco General Hospital Sleep Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No